CLINICAL TRIAL: NCT05125055
Title: Neoadjuvant Toripalimab and Albumin Paclitaxel /Cisplatin Versus Docetaxel/ Cisplatin/ 5-fluorouracil (TPF) on Pathological Response in Patients With Locally Advanced and Resectable Oral Squamous Cell Carcinoma
Brief Title: Neoadjuvant Anti-PD-1 and TP Versus TPF on Pathological Response in OSCC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Illuminate-2
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Oral Squamous Cell Carcinoma; Neoadjvant Therapy; Anti-PD-1; Chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab; Cisplatin; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant TTP (Experimental): The participants will receive two cycles of intravenous Albumin paclitaxel (260mg/ m^2), Cisplatin (75mg/ m^2) and Toripalimab (anti-PD-1 inhibitor, 240 mg) on d1 and d22.
  Interventions: Drug: Toripalimab (anti-programmed death-1 inhibitor); Drug: Albumin paclitaxel; Drug: Cisplatin
- Neoadjuvant TPF (Active Comparator): The participants will receive two cycles of intravenous Docetaxel (75 mg/m^2) on d1 and d22, Cisplatin (75 mg/m^2) on d1 and d22, and 5-Fluorouracil (750 mg/m^2/day) for 5 days (d1-5 and d22-26), the interval is 16±1 days.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Toripalimab (anti-programmed death-1 inhibitor) — The participants will receive two cycles of Toripalimab, with 21 days each. 240mg of Toripalimab will be used intravenously on the first day of each cycle.
  Arms: Neoadjuvant TTP
Drug: Albumin paclitaxel — The participants will receive two cycles of Albumin paclitaxel, with 21 days each. 260mg/m^2 of Albumin paclitaxel will be used intravenously on the first day of each cycle.
  Arms: Neoadjuvant TTP
Drug: Cisplatin — The participants will receive two cycles of Cisplatin, with 21 days each. 75mg/m^2 of Cisplatin will be used intravenously on the first day of each cycle.
Drug: Docetaxel — The participants will receive two cycles of Docetaxel, with 21 days each. 75mg/m^2 of Docetaxel will be used intravenously on the first day of each cycle.
  Arms: Neoadjuvant TPF
Drug: 5-Fluorouracil — The participants will receive two cycles of 5-Fluorouracil, with 21 days each. 750mg/m^2/d of 5-Fluorouracil will be used as a 120-hour continuous intravenous infusion on days 1 through 5.
  Arms: Neoadjuvant TPF

SUMMARY:
To compare the pathological efficacy of neoadjuvant Toripalimab and Albumin paclitaxel /Cisplatin (TTP) with Docetaxel/ Cisplatin/ 5-flurouracil (TPF) for patients with locally advanced resectable oral squamous cell carcinoma (OSCC), and to determine the safety of neoadjuvant TTP. In order to explore a better protocol of neoadjuvant therapy to improve the efficacy in patients with locally advanced OSCC.

DETAILED DESCRIPTION:
In the previous "Illuminate" trial, neoadjuvant anti-programmed death-1 (PD-1) of Toripalimab and Albumin paclitaxel /Cisplatin (TTP) therapy was used in 20 patients with locally advanced and resectable oral squamous cell carcinoma (OSCC), and the neoadjuvant therapy was well-tolerated. The major pathologic response (MPR) rate was 60% (12/20), including 30% (6/20) pathological complete response (pCR). Furthermore, the MPR might transfer to survival benefit in the patients received neoadjuvant therapy. Therefore, in this randomized trial, we aimed to compare the pathological response of neoadjuvant TTP therapy versus TPF chemotherapy in the patients with locally advanced OSCC (Illuminate-2 trial). A total of 80 patients will be enrolled in this trial, and the primary endpoint is MPR rate. The neoadjuvant TTP arm will receive two cycles of intravenous Albumin paclitaxel (260mg/ m^2), Cisplatin (75mg/ m^2) and Toripalimab (anti-PD1 inhibitor, 240 mg) on d1 and d22, followed by the standard treatment of surgery and postoperative adjuvant therapy. The neoadjuvant TPF arm will received two cycles of intravenous Docetaxel (75mg/m^2), Cisplatin (75mg/m^2) on d1 (d22), and 5-Fu(750mg/m^2/day) for 5 days (d1-5 and d22-26), followed by the standard treatment of surgery and postoperative adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old
2. Gender: male and female
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0-2
4. Histopathological diagnosis of oral squamous cell carcinoma (including tongue, gums, cheek, floor of mouth, hard palate, and posterior molar region)
5. Primary tumor with a clinical stage of III/IVA (T1-2/N1-2/M0 or T3-4a/cN0-2/M0, AJCC2018)
6. Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
7. Blood routine: white blood cells (WBCs) >3,000/mm3, hemoglobin >8 g/L, platelets >80,000/mm3
8. Liver function: alanine amino transferase/aspartate amino transferase (ALAT/ASAT) <2.5 times the upper limit of normal and bilirubin <1.5 times the upper limit of normal
9. Renal function: Serum creatinine <1.5 times the upper limit of normal
10. Coagulation function: INR, PT, APTT<1.5 times the upper limit of normal
11. Signed the informed consent form

Exclusion Criteria:

1. Unresolved grade 2 [(Common Terminology Criteria for Adverse Events (CTCAE 5.0)] or higher toxic reactions caused by previous anticancer treatments
2. Known allergic reaction to any ingredients or excipients of the therapy
3. Known history of malignancy, unless been cured and no recurrence for 5 years
4. Known history of radiation to head and neck
5. Active severe clinical infection (> National Cancer Institute (NCI)-CTCAE version 5.0 grade 2 infection)
6. Obvious cardiovascular abnormalities [such as myocardial infarction, superior vena cava syndrome, grade 2 or higher heart disease diagnosed according to the New York Heart Association (NYHA) classification 3 months before enrollment]
7. Patients receiving immunology-based treatment for any reason
8. Patients with a history of active bleeding, coagulopathy, or receiving coumarin anticoagulation therapy
9. Pregnant or lactating women
10. Uncontrollable hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >90 mmHg) or cardiovascular diseases with clinical significance (such as activity), such as cerebrovascular accidents (≤ 6 months before screening), myocardial infarction (≤6 months before screening), unstable angina pectoris, NYHA grade II or above congestive heart failure, or severe arrhythmia that cannot be controlled by drugs or has a potential impact on trial treatment
11. Complicated with severe, uncontrolled infection or known human immunodeficiency virus (HIV) infection, or diagnosed as acquired immunodeficiency syndrome (AIDS); or uncontrolled autoimmune disease; or history of allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or solid organ transplantation
12. Participation in other clinical trials within 30 days before enrollment
13. Other situations that the investigator considers unsuitable with respect to participating in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 3 months
  The major pathologic response (MPR): the percentage of tumor cells before and after treatment was compared according to biopsy specimens before neoadjuvant therapy and pathological specimens after surgery; the percentage of residual viable tumor (RVT) cells was evaluated on resected tumor slides. MPR was defined as ≤ 10% RVT%.

SECONDARY OUTCOMES:
2-year disease-free survival rate | 24 months
  Disease-free survival was calculated from the date of randomization to tumor recurrence or death from any cause.
2-year overall survival rate | 24 months
  Overall survival was calculated from the date of randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the primary study report might be shared depending on the condition of trial completion.
Supporting Information: Study Protocol, SAP, ICF